CLINICAL TRIAL: NCT00002720
Title: QUADRANTECTOMY PLUS AXILLARY DISSECTION VERSUS QUADRANTECTOMY ALONE IN MAMMOGRAPHIC STAGE T1N0 BREAST CANCER PATIENTS AGED OVER 65 YEARS
Brief Title: Surgery With or Without Lymph Node Removal in Treating Older Women With Stage I Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064573; CNR-9502; EU-95020
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2000-08

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

INTERVENTIONS:
Drug: tamoxifen citrate
Procedure: conventional surgery

SUMMARY:
RATIONALE: Surgery to remove axillary lymph nodes may be an effective treatment for women with breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of therapy with or without axillary lymph node dissection following quadrantectomy in treating older women with stage I breast cancer that is estrogen receptor positive.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of quadrantectomy with or without axillary lymph node dissection, followed by tamoxifen in terms of local and distant relapse rates and overall survival of patients with stage I, invasive breast cancer.
* Determine the relationship between biological variables, such as hormone receptor status, cell proliferation, and DNA ploidy, and the clinical outcome of the disease in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo quadrantectomy with dissection of level I and II axillary lymph nodes.
* Arm II: Patients undergo quadrantectomy without axillary lymph node dissection. Patients on both arms receive tamoxifen daily for 5 years.

Patients are followed every 4 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 642 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage I, invasive breast cancer
* Hormone receptor status:

  * Estrogen receptor positive
  * Progesterone receptor positive or negative

PATIENT CHARACTERISTICS:

Age:

* 65 to 80

Sex:

* Female

Menopausal status:

* Postmenopausal

Performance status:

* Not specified

Life Expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No serious disease that would preclude surgery
* No other prior or concurrent malignancy except basal cell carcinoma or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 642 (Estimated)
Dates: Start 1995-12; Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Martelli, MD, Study Chair — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Istituto Nazionale per lo Studio e la Cura dei Tumori, Milano (Milan), Italy

REFERENCES:
- [Derived] Martelli G, Boracchi P, Ardoino I, Lozza L, Bohm S, Vetrella G, Agresti R. Axillary dissection versus no axillary dissection in older patients with T1N0 breast cancer: 15-year results of a randomized controlled trial. Ann Surg. 2012 Dec;256(6):920-4. doi: 10.1097/SLA.0b013e31827660a8. PMID 23154393